CLINICAL TRIAL: NCT03134508
Title: Evaluation of Adherence to Guidelines, and of the Risk to Benefit Ratio, in the Use of TNFα Antagonists in Pregnant Women With Inflammatory Bowel Diseases. Study on the French National PMSI Database
Brief Title: Population Based Evaluation of the Use of TNFα Antagonists in Pregnant Women With Inflammatory Bowel Diseases
Acronym: EVASION
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LUU AOI 2016
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant IBD women treated: pregnant IBD women treated by antiTNFα
  Interventions: Other: treated by antiTNFα
- pregnant IBD women not treated: pregnant IBD women not treated by antiTNFα
  Interventions: Other: not treated by antiTNFα

INTERVENTIONS:
Other: treated by antiTNFα — pregnant IBD women treated by antiTNFα
  Groups: pregnant IBD women treated
Other: not treated by antiTNFα — pregnant IBD women not treated by antiTNFα
  Groups: pregnant IBD women not treated

SUMMARY:
: Inflammatory bowel diseases (IBD), such as Crohn's disease (CD) and ulcerative colitis (UC) need long term treatments which can conflict with a desire of pregnancy in women. Uncontrolled IBD increases the risk of poor pregnancy outcomes [1]. Antitumor Necrosis Factor α (antiTNFα) are commonly used, off-label, in pregnancy but with the risk of treatment-related complications. Existing recommendations on the use of antiTNFα during pregnancy are conflicting and only rely on expert opinions. This study was aimed to assess appropriateness and risk to benefit ratio of antiTNFα treatment during pregnancy in women with IBD, for both the mother and the baby until the end of the first year.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy between 01/01/2011 and 31/12/2014
* Diagnosis of IBD (Crohn's disease or Ulcerative Colitis)

Exclusion Criteria:

* Non IBD indication of antiTNFα treatment

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women with a diagnosis of IBD
Sampling Method: Probability Sample
Enrollment: 8726 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Overall complications | 9 months
  composite criteria composed by:
  * Disease related complications
  * Treatment related complications
  * Pregnancy related complications

SECONDARY OUTCOMES:
Infectious Complications in the children born from IBD mothers | The first year of life
  Occurrence of infectious complications during the first year of life

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Dijon, Dijon, France